CLINICAL TRIAL: NCT03065764
Title: 89Zirconium-labeled Pembrolizumab as Predictive Imaging Biomarker of Response and Toxicity in Pembrolizumab Treated Patients With Non-small-cell Lung Cancer - a Feasibility Study
Brief Title: 89Zr-labeled Pembrolizumab in Patients With Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. dr. E.F. Smit, Prof. dr. E.F. Smit, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PN221
Record Dates: First submitted 2017-01-20; First posted 2017-02-28 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Pembrolizumab; 89Zirconium
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Other): For the first 3 patients, PET scans will be obtained at 1, 72 and 120 hours post tracer injection to determine the optimal scan time point and to perform biodistribution measurements and dosimetry. All subsequent 7 patients receive only 1 PET scan post-injection (i.e. two PET scans).
  Interventions: Drug: 89Zr-Pembrolizumab

INTERVENTIONS:
Drug: 89Zr-Pembrolizumab — eligible subjects will undergo two whole body immuno-PET scans with a non-therapeutic tracer dose (2 mg) of 89Zr-pembrolizumab; one with and one without a preceding "cold" therapeutic dose of pembrolizumab.
  Other Names: Pembrolizumab

SUMMARY:
After a screening phase of up to 42 days, eligible subjects will undergo two whole body immuno-PET scans with a non-therapeutic tracer dose (2 mg) of 89Zr-pembrolizumab; one with and one without a preceding "cold" therapeutic dose of pembrolizumab. For the first 3 patients, PET scans will be obtained at 1, 72 and 120 hours post tracer injection to determine the optimal scan time point and to perform biodistribution measurements and dosimetry. All subsequent patients receive only 1 PET scan post-injection (i.e. two PET scans). The optimal time point is expected to be at day 5 post-injection. Pembrolizumab treatment will continue every three weeks until two years of therapy have been administered, disease progression, or unacceptable adverse event(s).

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of stage IV, EGFR wt and EML4/ALK fusion negative NCSLC and have received at least one line of platinum based doublet chemotherapy and disease progression by RECIST 1.1 on the last systemic treatment.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be 18 years of age, or above on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Must provide newly obtained tissue from a core or excisional biopsy of a tumor lesion and are willing to undergo a second biopsy when the 89Zr-pembrolizumab PET scan shows heterogeneous uptake.
6. Have a performance status of 0-2 on the ECOG Performance Scale.
7. Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation (day 12).
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy in a dose higher than the equivalent of 10 mg prednisolone once daily or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with asymptomatic CNS metastases are allowed to enter the study. Subjects with previously treated brain metastases may participate provided they are stable and are not using steroids for at least 7 days prior to trial treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has received > 30 Gy of thoracic radiotherapy within 6 months of starting Pembrolizumab.
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events of 89Zr-pembrolizumab will be assessed by CTCAE v 4.0. | up to 2 years
  Safety assessment will be measured through adverse events, changes in laboratory test results, changes in vital signs, and exposure to 89Zr-pembrolizumab. Adverse event data will be recorded and summarized according to NCI CTCAE v4.0.
Description of 89Zr-pembrolizumab uptake in tumor lesions by measuring standardized uptake value (SUV) on the 89Zr-pembrolizumab-PET scans | up to 2 years
  Description of 89Zr-pembrolizumab uptake in tumor lesions by measuring standardized uptake value (SUV) on the 89Zr-pembrolizumab-PET scans
Visual 89Zr-pembrolizumab uptake in tumor lesions will be scored as positive or negative. | up to 2 years
  Visual 89Zr-pembrolizumab uptake in tumor lesions will be scored as positive or negative.
Characterize tumor uptake heterogeneity between patients and within and between tumor lesions of the same patient | up to 2 years
  Intrapatient and interpatient 89Zr-pembrolizumab tumor uptake heterogeneity is expected and can be visualized.

SECONDARY OUTCOMES:
Characterize the relationship between 89Zr-pembrolizumab tumor uptake and tumor and TIL PD-1 and PD-L1 expression as well as other blood and tissue parameters | up to 2 years
  Differences in 89Zr-pembrolizumab tumor uptake can be explained by (spatial) differences in tumor and TIL PD-1 and PD-L1 expression.
Explore the relationship between 89Zr-pembrolizumab organ uptake with irAEs. The focus will be on the gut, lung, liver, thyroid and pituitary. | up to 2 years
  The level of tracer uptake in target irAE tissues correlates with immune-related toxicity.
Assess uptake of 89Zr-pembrolizumab in normal tissues by measuring standardized uptake value (SUV) to evaluate the biodistribution and dosimetry. | up to 2 years
  Assess uptake of 89Zr-pembrolizumab in normal tissues by measuring standardized uptake value (SUV) to evaluate the biodistribution and dosimetry.

CONTACTS AND LOCATIONS:
Overall Officials: EF Smit, Principal Investigator — VUMedicalcentre
Locations (1):
- VUMedicalCentre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No